CLINICAL TRIAL: NCT00793598
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study of the Safety, Tolerability and Population Pharmacokinetics of CMX001 in Post-Transplant Subjects With BK Virus Viruria
Brief Title: CMX001 in Post-transplant Patients With BK Virus Viruria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMX001-104
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Viruria
Keywords: CMX001; Kidney transplant; HSCT transplant; BK Virus; Post kidney transplant patients with BK virus viruria > 10^4; Post HSCT transplant patients with BK virus viruria > 10^4
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brincidofovir (Experimental): Under Amendments 1 and 2, subjects received 1 of 2 dose regimens of brincidofovir, as follows:
  * 20 mg BCV once weekly (QW) on Days 0, 7, and 14; or
  * 10 mg BCV twice weekly (BIW) BIW on Days 0, 3, 7, 10, and 14.
  Under Amendment 3, subjects received 40 mg BCV QW for a total of 5 doses on Days 0, 7, 14, 21, and 28.
  Interventions: Drug: Brincidofovir
- Placebo (Placebo Comparator): Under Amendments 1 and 2, subjects received placebo twice weekly (BIW) for a total of 5 doses on Days 0, 3, 7, 10, and 14.
  Under Amendment 3, subjects received placebo once weekly (QW) for a total of 5 doses on Days 0, 7, 14, 21, and 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Brincidofovir
  Other Names: BCV; CMX001
  Arms: Brincidofovir

SUMMARY:
This was a randomized, double-blind, multiple-dose placebo-controlled study of oral brincidofovir (BCV) in hematopoietic stem cell transplant and renal transplant recipients with BK virus viruria.

DETAILED DESCRIPTION:
This was a randomized, double-blind, multiple-dose placebo-controlled study of oral brincidofovir (BCV) in hematopoietic stem cell transplant and renal transplant recipients with BK virus infection.

Subjects received blinded study medication for a total of 5 doses in 1 of the following regimens:

* 10 mg BCV administered twice weekly (BIW) on Days 0, 3, 7, 10, 14.
* 20 mg BCV administered once weekly (QW) on Days 0, 7, and 14 and placebo administered on Days 3 or 10.
* Placebo administered BIW on Days 0, 3, 7, 10 ,14.
* 40 mg BCV administered QW on Days 0, 7, 14, 21, and 28.
* Placebo administered QW on Days 0, 7, 14, 21, and 28.

ELIGIBILITY:
Inclusion Criteria:

For inclusion into the trial, subjects were required to fulfill all of the following criteria:

1. Aged between 18 to 75 years, inclusive. Males must have been able and willing to use adequate contraceptive methods throughout the study and for 3 months after the final dose. Females must have been post-menopausal, surgically sterile, or willing to use adequate contraception for the duration of the study (screening through the Day 48 visit).
2. Were renal or hematopoietic stem cell transplant patients who met the following criteria:

   1. Renal transplant patients who:

      * Were at least 28 days post transplant;
      * Were in stable condition with hemoglobin >10 g/100 mL;
      * Had no evidence of graft rejection (i.e., serum creatinine was not increasing [±30%], creatinine clearance was not decreasing);
      * Were on a stable immunosuppressant regimen for at least 14 days prior to dosing.
      * Had either urine levels of BK virus DNA ≥10^4 copies/mL without viremia or plasma levels of BK virus DNA <10^4 copies/mL (with or without viruria).
   2. Stem cell transplant patients who:

      * Were a minimum of 3 days post documentation of successful engraftment as evidenced by an absolute neutrophil count >500 cells/mm3;
      * Had urine levels of BKV ≥10^4 copies/mL.
3. Had GFR >30 mL/min.
4. Were able to swallow tablets.
5. Were willing and able to understand and provide written informed consent.
6. Were willing and able to participate in all required study activities for the duration of the study (including ingestion of oral medication).

Exclusion Criteria

Any of the following was regarded as a criterion for exclusion from the trial:

1. Females who were currently nursing or pregnant.
2. Were using illicit drugs or abusing alcohol.
3. Had hypersensitivity to cidofovir or brincidofovir.
4. Had received aminoglycosides (intravenously) or NSAIDS (except as given for cardioprotective treatment) within 7 days prior to enrollment; had received leflunomide, cidofovir, or any other medication for treatment of BK virus infection or disease within 14 days prior to enrollment; had received any investigational drug (including maribavir) within 30 days prior to enrollment.
5. Were HIV positive (results must have been obtained within 1 year prior to dosing); had active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection as evidenced by plasma levels of HCV RNA or HBV DNA, respectively.
6. Were renal transplant patients with evidence of biopsy proven acute rejection in the 3 weeks prior to enrollment. This exclusion criterion applied only to those patients for whom a biopsy was performed within the 3 weeks prior to enrollment.
7. Were stem cell transplant patients who:

   1. Had cystitis ≥Grade 3 National Cancer Institute, Common Terminology Criteria for Adverse Events version 3.0.
   2. Had Grade 3 or 4 graft versus host disease (GVHD).
   3. Had untreated or uncontrolled Grade 2 GVHD.
   4. Had received ganciclovir or valganciclovir within 14 days prior to enrollment.
8. Had mucositis that prevented ingestion of oral medication.
9. Had hypotony, uveitis, or retinitis or any intraocular pathology that would have predisposed the patient to any one of these conditions.
10. Had unstable or poorly controlled diabetes, defined as having frequent hypoglycemic and/or hyperglycemic events on a daily basis (brittle diabetes), with fluctuating short acting insulin requirements daily, or requiring unpredictable insulin supplementation to oral hypoglycemic agents on a regular basis.
11. Had bilirubin >2.5 x the upper limit of normal.
12. Had cardiovascular disease which, in the opinion of the investigator, would have interfered with the conduct of the study.
13. Had any of the following autoimmune diseases: Addison's disease, autoimmune hemolytic anemia, autoimmune hepatitis, bullous pemphigoid, celiac disease, dermatomyositis, active Goodpasture's syndrome, idiopathic thrombocytopenic purpura, active lupus erythematosus, multiple sclerosis, myasthenia gravis, pemphigus vulgaris, polymyositis, primary biliary cirrhosis, vasculitis, Wegener's granulomatosis.
14. Had active malignancies (with the exception of basal cell carcinoma or the condition under treatment for hematopoietic stem cell transplant patients).
15. Had concurrent or ongoing ≥Grade 2 gastrointestinal symptoms including nausea, vomiting, diarrhea, constipation, or gastroenteritis. Patients with active gastrointestinal disease including inflammatory bowel disease, irritable bowel syndrome, or celiac sprue.
16. Had any other condition including abnormal laboratory values that would have, in the judgement of the investigator, put the subject at increased risk for participating in the trial, or interfered with the conduct of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Tulane Center for Abdominal Transplant, New Orleans, Louisiana
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mt. Sinai Medical Center, New York, New York
  - UNC Kidney Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Vermont, Burlington, Vermont
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 HCT subject in the 40 mg BCV QW treatment arm was not dosed with BCV and, therefore, is not included in further analyses.
Groups:
- 10 mg BCV BIW RT: Renal transplant (RT) recipients who received 10 mg brincidofovir (BCV) administered twice weekly (BIW) on Days 0, 3, 7, 10, and 14.
- 10 mg BCV BIW HCT: Hematopoietic stem cell transplant (HCT) recipients who received 10 mg brincidofovir (BCV) administered twice weekly (BIW) on Days 0, 3, 7, 10, and 14.
- 20 mg BCV QW HCT: Hematopoietic stem cell transplant (HCT) recipients who received 20 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, and 14.
- Placebo BIW HCT: Hematopoietic stem cell transplant (HCT) recipients who received placebo twice weekly (BIW) under Amendment 2.
- 40 mg BCV QW RT: Renal transplant (RT) recipients who received 40 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, 14, 21, and 28.
- 40 mg BCV QW HCT: Hematopoietic stem cell transplant (HCT) recipients who received 40 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, 14, 21, and 28.
- Placebo QW RT: Renal transplant (RT) recipients who received placebo once weekly (QW) under Amendment 3.
- Placebo QW HCT: Hematopoietic stem cell transplant (HCT) recipients who received placebo once weekly (QW) under Amendment 3.
Period: Overall Study
Arm/Group | 10 mg BCV BIW RT | 10 mg BCV BIW HCT | 20 mg BCV QW HCT | Placebo BIW HCT | 40 mg BCV QW RT | 40 mg BCV QW HCT | Placebo QW RT | Placebo QW HCT
Started | 1 | 1 | 1 | 2 | 8 | 8 | 4 | 4
Completed | 1 | 0 | 1 | 2 | 8 | 7 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Patient Request | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Subject not dosed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 HCT subject in the 40 mg BCV QW treatment arm was not dosed with BCV and, therefore, is not included in this analysis.
Groups:
- 10 mg BCV BIW: Subjects who received 10 mg brincidofovir (BCV) administered twice weekly (BIW) on Days 0, 3, 7, 10, and 14.
- 20 mg BCV QW: Subjects who received 20 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, and 14.
- Placebo BIW: Subjects who received placebo twice weekly (BIW) under Amendment 2.
- 40 mg BCV QW: Subjects who received 40 mg brincidofovir (BCV) administered once weekly (QW) on Days 0 7, 14, 21, and 28.
- Placebo QW: Subjects who received placebo once weekly (QW) under Amendment 3.
- Total: Total of all reporting groups
Arm/Group | 10 mg BCV BIW | 20 mg BCV QW | Placebo BIW | 40 mg BCV QW | Placebo QW | Total
Number analyzed (Participants) | 2 | 1 | 2 | 15 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 60 (0) | 60 (2) | 55.5 (15.14) | 51.0 (10.46) | 51.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 3 | 4 | 8
  Male | 2 | 1 | 1 | 12 | 4 | 20
Type of transplant received [Count of Participants; unit: Participants]
  Hematopoietic stem cell transplant recipients | 1 | 1 | 2 | 7 | 4 | 15
  Renal transplant recipients | 1 | 0 | 0 | 8 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events in Post-Transplant Patients With BK Virus Viruria
Description: The primary objective of this study was to determine the safety and tolerability of brincidofovir (BCV) in post-transplant patients with BK virus viruria. Safety measures included adverse events, clinical laboratory values, vital signs, and renal and gastrointestinal function.
Time Frame: 35 days (Day 0 to Day 35)
Population: 1 subject in the 40 mg BCV QW HCT treatment arm was not dosed with BCV and, therefore, was not included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg BCV BIW RT: Renal transplant (RT) recipients who received 10 mg brincidofovir (BCV) administered twice weekly
- 20 mg BCV BIW HCT: Hematopoietic stem cell transplant (HCT) recipients who received 20 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, and 14.
Arm/Group | 10 mg BCV BIW RT | 10 mg BCV BIW HCT | 20 mg BCV BIW HCT | Placebo BIW HCT | 40 mg BCV QW RT | 40 mg BCV QW HCT | Placebo QW RT | Placebo QW HCT
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 8 | 7 | 4 | 4
Participants
  Subjects who experienced at least 1 an adverse event | 1 | 1 | 1 | 2 | 8 | 7 | 3 | 4
  Subjects who did not experience an adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Percentage of Patients Who Achieved BK Viruria Resolution
Description: The percentage of subjects who cleared the virus was calculated. Concentrations below the lower limit of quantification were indicated as below the limit of quantitation and were considered "cleared".
Time Frame: 28 days
Population: Hematopoietic stem cell (HCT) recipients and renal transplant (RT) recipients enrolled under Amendment 3 who had detectable BK viruria at baseline (Day 0). 1 HCT subject in the 40 mg BCV QW treatment arm was not dosed with BCV and, therefore, is not included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 40 mg BCV QW: Subjects who received 40 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, 14, 21, and 28.
- Placebo: Subjects who received placebo once weekly (QW) on Days 0, 7, 14, 21 and 28.
Arm/Group | 40 mg BCV QW | Placebo
Number analyzed (Participants) | 15 | 8
Participants
  HCT recipients: number analyzed (Participants) | 7 | 4
  HCT recipients: Subjects who cleared viruria | 1 | 0
  HCT recipients: Subjects who did not clear viruria | 6 | 4
  RT Recipients: number analyzed (Participants) | 8 | 4
  RT Recipients: Subjects who cleared viruria | 1 | 0
  RT Recipients: Subjects who did not clear viruria | 7 | 4

3. Secondary Outcome: Number of Patients Who Achieved a Clinically Significant Decrease in BK Viruria
Description: A 2-log drop in viruria or viremia or clearance of virus was considered significant. Percentages of subjects with a 2-log drop in viral load were calculated.
Time Frame: 28 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 40 mg BCV QW: Subjects randomized to receive 40 mg brincidofovir (BCV) administered once weekly (QW) on Days 0, 7, 14, 21, and 28.
- Placebo QW: Subjects who received placebo once weekly (QW) on Days 0, 7, 14, 21 and 28.
Arm/Group | 40 mg BCV QW | Placebo QW
Number analyzed (Participants) | 15 | 8
Participants
  HCT recipients: number analyzed (Participants) | 7 | 4
  HCT recipients: Subjects with 2-log drop from Day 0 | 1 | 1
  HCT recipients: Subjects without 2-log drop from Day 0 | 6 | 3
  RT Recipients: number analyzed (Participants) | 8 | 4
  RT Recipients: Subjects with 2-log drop from Day 0 | 0 | 0
  RT Recipients: Subjects without 2-log drop from Day 0 | 8 | 4

ADVERSE EVENTS:
Time Frame: Day 0 to Day 35
Description: 1 HCT subject in the 40 mg BCV QW treatment arm was not dosed with BCV and, therefore, is not included in this analysis.
Arm/Group | 10 mg BCV BIW RT | 10 mg BCV BIW HCT | 20 mg BCV QW HCT | Placebo BIW HCT | 40 mg BCV QW RT | 40 mg BCV QW HCT | Placebo QW RT | Placebo QW HCT
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/2 | 0/8 | 2/7 | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 2/2 | 8/8 | 7/7 | 3/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg BCV BIW RT (N=1) | 10 mg BCV BIW HCT (N=1) | 20 mg BCV QW HCT (N=1) | Placebo BIW HCT (N=2) | 40 mg BCV QW RT (N=8) | 40 mg BCV QW HCT (N=7) | Placebo QW RT (N=4) | Placebo QW HCT (N=4)
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute graft versus host disease skin (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreas transplant rejection (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg BCV BIW RT (N=1) | 10 mg BCV BIW HCT (N=1) | 20 mg BCV QW HCT (N=1) | Placebo BIW HCT (N=2) | 40 mg BCV QW RT (N=8) | 40 mg BCV QW HCT (N=7) | Placebo QW RT (N=4) | Placebo QW HCT (N=4)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood amylase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Androgen deficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment.